CLINICAL TRIAL: NCT02732899
Title: Sirolimus in Conjunction With EYLEA® (Aflibercept) Versus EYLEA® Alone for Exudative AMD
Brief Title: Sirolimus in Conjunction With Eylea vs Eylea Alone for Exudative AMD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maturi, Raj K., M.D., P.C. (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RKM009
Record Dates: First submitted 2016-04-05; First posted 2016-04-11 (Estimated); Results first posted 2018-02-14 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-01

CONDITIONS: Exudative Age Related Macular Degeneration
Keywords: AMD
MeSH Terms: interventions — Sirolimus; aflibercept

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Sirolimus 440ug for intravitreal injection will be provided in sterile single-use glass vials. One single-dose vial will be packaged in a box for each patient injection. Sirolimus injections will be given at baseline, week 4, 12, 20 and 28. EYLEA® (aflibercept) intravitreal injections will be given at week 1, 8, 16, 24 and 32.
  Interventions: Drug: Sirolimus; Drug: EYLEA
- Group 2 (Active Comparator): Intravitreal injection of EYLEA® (aflibercept) will be given at baseline, week 8, 16, 24 and 32. Sham injections will be given at week 1, 4, 12, 20, and 28 in order to maintain masking of patient to treatment assignment
  Interventions: Drug: EYLEA

INTERVENTIONS:
Drug: Sirolimus
  Other Names: DE-109
  Arms: Group 1
Drug: EYLEA
  Other Names: aflibercept

SUMMARY:
To determine safety and efficacy of intravitreal injections of Sirolimus with adjunct EYLEA in subjects with exudative age related macular degeneration (AMD) with persistent intraretinal or subretinal edema due to neovascular AMD despite previous intravitreal anti-vascular endothelial growth factor (antiVEGF) treatment.

DETAILED DESCRIPTION:
This study is a single-center, masked, randomized, 36 week study, designed to evaluate the safety and treatment efficacy of intravitreal Sirolimus with adjunct EYLEA® (aflibercept) in patients with persistent edema due to neovascular AMD versus EYLEA® (aflibercept) alone. Twenty (20) patients will be randomized to receive study medication in a 1:1 ratio. Study treatment will be administered by intravitreal injections. The sham injections given in the EYLEA® alone group are needleless and they are given in order to help preserve the masking of those subjects in that treatment group.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, 50 years of age or older at baseline
2. Patient has completed/signed an informed consent prior to any study-related procedures and is able to follow study instructions and likely to complete all required visits.

   • Ocular Inclusion Criteria (Study eye only):
3. BCVA 5 - 75 (20/800-20/30), inclusive, in study eye; if both eyes are eligible, the eye with the best potential visual improvement as determined by the investigator will be selected for treatment.
4. Presence of choroidal neovascularization secondary to AMD
5. At least 3 previous intravitreal anti-VEGF injections in the past 6 months
6. Injection of antiVEGF may be deferred for at least 4 weeks from randomization based on clinical assessment of AMD by the investigator.
7. Clear ocular media and adequate pupil dilation to permit good quality photographic imaging -

Exclusion Criteria:

1. Females who are pregnant, nursing, planning a pregnancy or who are of childbearing potential not using a reliable method of contraception.
2. History or current evidence of hypersensitivity to any components of the study medication or fluorescein, as assessed by the investigator.
3. Participation in any investigational drug or device study within 30 days prior to baseline
4. History or current evidence of a medical condition that may, in the opinion of the investigator, preclude the safe administration of study medication or affect the results of the study.

   • Ocular Exclusion Criteria (Study eye only):
5. Decrease of greater than 150 microns in central subfield thickness as measured by OCT since the last intravitreal injection in the study eye
6. Aphakia
7. History of pars plana vitrectomy in the study eye
8. History of major ophthalmic surgery in the study eye in the past 3 months and any ophthalmic surgery in the study eye within the past 30 days
9. History of significant ocular disease or condition other than exudative AMD that may confound results
10. Uncontrolled glaucoma (defined as intraocular pressure >21mm Hg despite treatment with two or more ocular hypotensive medications at baseline)
11. No active ocular or periocular infections, or ocular malignancy including lymphoma
12. Presence of significant epiretinal membrane
13. Significant vitreoretinal traction

    -

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-04; Primary Completion 2017-03-20 (Actual); Study Completion 2017-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raj K Maturi, MD, Principal Investigator — Raj K. Maturi, MD, PC
Locations (1):
- Raj K Maturi MD PC, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rowe LW, Minturn RJ, Burgett LA, Bracha P, Maturi RK. Intravitreal sirolimus with adjunct aflibercept versus aflibercept monotherapy for persistent, exudative age-related macular degeneration: a pilot study. Int J Retina Vitreous. 2023 Jan 5;9(1):1. doi: 10.1186/s40942-022-00437-6. PMID 36604756

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Sirolimus 440ug for intravitreal injection will be provided in sterile single-use glass vials. One single-dose vial will be packaged in a box for each patient injection. Sirolimus injections will be given at baseline, week 4, 12, 20 and 28. EYLEA® (aflibercept) intravitreal injections will be given at week 1, 8, 16, 24 and 32.
  Sirolimus
  EYLEA
- Group 2: Intravitreal injection of EYLEA® (aflibercept) will be given at baseline, week 8, 16, 24 and 32. Sham injections will be given at week 1, 4, 12, 20, and 28 in order to maintain masking of patient to treatment assignment
  EYLEA
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Full Range); unit: years] | 71 [69 to 90] | 77 [63 to 91] | 74 [63 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 10 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Central Subfield Thickness on OCT From Baseline to Week 36
Description: the amount of change in intraretinal and subretinal fluid as measured by microns of central subfield thickness (CST) on Heidelberg Optical Coherence Tomography (OCT)
Time Frame: baseline to week 36
Measure: Mean (Full Range); unit: microns
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 10 | 10
microns | -54 [-74 to -34] | -.1 [-.6 to 0.5]

2. Secondary Outcome: Change in Best Corrected Visual Acuity (BCVA) From Baseline to Week 36
Time Frame: baseline to week 36
Measure: Mean (Full Range); unit: letters
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 10 | 10
letters | 2.5 [1.6 to 3.8] | 0.8 [0.444 to 2.2]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 3/10 | 0/10
Other Adverse Events (participants affected / at risk) | 10/10 | 5/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=10) | Group 2 (N=10)
worsening hypertension (Vascular disorders) | 1 (1) | 0 (0)
pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=10) | Group 2 (N=10)
worsening subretinal hemorrhage (Eye disorders) | 0 (0) | 1 (1)
progressed posterior capsule opacification (Eye disorders) | 2 (2) | 0 (0)
urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0)
sinusitis (Infections and infestations) | 1 (1) | 0 (0)
dot hemorrhage on retina (Eye disorders) | 2 (2) | 0 (0)
progressed nuclear sclerotic cataract (Eye disorders) | 1 (1) | 0 (0)
subretinal hemorrhage (Eye disorders) | 0 (0) | 1 (1)
bronchitis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
hyperemia (Eye disorders) | 2 (2) | 0 (0)
increased metemorphopsia (Eye disorders) | 2 (3) | 0 (0)
foreign body sensation (Eye disorders) | 1 (1) | 0 (0)
eye pain (Eye disorders) | 1 (2) | 1 (1)
tooth infection (Infections and infestations) | 1 (1) | 0 (0)
chalazion (Eye disorders) | 0 (0) | 1 (1)
combigan allergy (General disorders) | 1 (1) | 0 (0)
epiphora (Eye disorders) | 0 (0) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
eyelid edema (Eye disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-11): https://cdn.clinicaltrials.gov/large-docs/99/NCT02732899/Prot_SAP_000.pdf